CLINICAL TRIAL: NCT07329400
Title: Turkish Adaptation of the Burnt Hand Outcome Tool (BHOT): A Validity and Reliability Study in Adult Patients With Hand Burns
Brief Title: Turkish Adaptation and Validation of the Burnt Hand Outcome Tool (BHOT)
Status: Recruiting | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Collaborators: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Pariya Pouriyamanesh, MSc student in Physiotherapy and Rehabilitation, Necmettin Erbakan University
Other Study IDs: NecmettinEU-FTR-PP-01
Record Dates: First submitted 2025-11-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hand Burn; Hand Injuries; Burn Injuries
Keywords: Hand Burns; Burnt Hand Outcome Tool (BHOT); Validation Study; Reproducibility of Results; Burn Injuries
MeSH Terms: conditions — Hand Injuries; Burns

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Burnt Hand Outcome Tool (BHOT) - Turkish Version — Assessment using the Turkish version of the Burnt Hand Outcome Tool (BHOT) for validity and reliability evaluation; no treatment is applied.

SUMMARY:
The goal of this observational study is to evaluate the validity and reliability of the Turkish adaptation of the Burnt Hand Outcome Tool (BHOT) in adults with a history of hand burns. The participant population will include adults aged 18 years and older who have experienced unilateral or bilateral hand burns and can read and understand Turkish.The main questions this study aims to answer are:

Does the Turkish version of the BHOT demonstrate high internal consistency, test-retest reliability, and construct validity? How strongly are BHOT scores associated with objective hand function measures such as grip strength and sensory evaluation? Participants will not be assigned to comparison groups, as this is a methodological validation study.

Participants will: Complete a sociodemographic information form. Complete the Turkish version of the BHOT and the QuickDASH questionnaire. Undergo objective assessments including hand grip strength using a dynamometer and sensory evaluation using Semmes-Weinstein monofilaments. Participate in repeated assessments at baseline, 1 month, 3 months and 6 months for reliability analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* History of second-degree or higher burn injury in one or both hands
* Ability to read and understand Turkish
* Willingness to participate and provision of written informed consent

Exclusion Criteria:

* History of trauma, surgery, or rheumatologic disease affecting hand function prior to the burn injury
* Age under 18 years
* Cognitive impairment or psychiatric disorder preventing completion of the questionnaires
* Refusal to participate or withdrawal from the study at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years and older with a history of second-degree or higher burn injury in one or both hands who are receiving outpatient or inpatient care at the burn unit. All participants are able to read and understand Turkish and provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Reliability of the Turkish Version of the Burnt Hand Outcome Tool (BHOT) | Baseline , 1 month, 3 months, and 6 months
  Total score of the Turkish version of the Burnt Hand Outcome Tool (BHOT-T), a patient-reported outcome measure assessing functional, aesthetic, sensory, and psychosocial outcomes in adults with hand burns. The BHOT-T consists of 20 items, each scored on a Likert scale.
  Total scores range from 0 to 80, with higher scores indicating worse outcomes / greater negative impact of hand burns on hand function and quality of life.
Construct Validity of Burnt Hand Outcome Tool-Turkish | baseline, 1 month, 3 months, and 6 months
  Construct validity will be assessed using confirmatory factor analysis (CFA) to evaluate the factor structure of the Turkish version of Burnt Hand Outcome Tool.

SECONDARY OUTCOMES:
Convergent Validity With QuickDASH | Baseline, 1 month, 3 months, and 6 months
  Total score of the Quick Disabilities of the Arm, Shoulder and Hand questionnaire (Quick DASH), a patient reported outcome measure assessing upper extremity disability. Scores are reported as units on a scale from 0 to 100, with higher scores indicating greater disability.
Hand Grip Strength | Baseline
  Hand grip strength measured in kilograms (kg) using a hand dynamometer in adults with hand burns.
Sensory Function Assessment | Baseline
  Sensory function of the hand assessed using the Semmes-Weinstein Monofilament Test, reported as monofilament level indicating cutaneous sensory threshold.
Discriminant Validity by Clinical Characteristics | Baseline
  Discriminant validity will be evaluated by comparing total scores of the Turkish version of the Burnt Hand Outcome Tool (Burnt Hand Outcome Tool - Turkish version, BHOT-T) across predefined clinical subgroups, including burn severity, history of skin grafting, and working status.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital (Konya Şehir Hastanesi), Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No